CLINICAL TRIAL: NCT02757755
Title: Ascending Dose Study of the Safety of AB-SA01 When Topically Applied to Intact Skin of Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double
Other Study IDs: AB-SA01-01; WRAIR-2285 (Other: Walter Reed Army Institute of Research)
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 10^8 (Experimental): AB-SA01 (10^8) and Placebo
  Interventions: Biological: AB-SA01 (10^8 PFU per phage); Biological: Placebo (for Cohort 10^8)
- Cohort 10^9 (Experimental): AB-SA01 (10^9) and Placebo
  Interventions: Biological: AB-SA01 (10^9 PFU per phage); Biological: Placebo (for Cohort 10^9)

INTERVENTIONS:
Biological: AB-SA01 (10^8 PFU per phage) — Gauze pads will be saturated with AB-SA01 and then applied to each subject's volar forearm and covered with occlusive dressing once daily for 3 consecutive days. Placement of the gauze to each subject's right or left volar forearm will be randomized and double-blinded.
  Arms: Cohort 10^8
Biological: AB-SA01 (10^9 PFU per phage) — Gauze pads will be saturated with AB-SA01 and then applied to each subject's volar forearm and covered with occlusive dressing once daily for 3 consecutive days. Placement of the gauze to each subject's right or left volar forearm will be randomized and double-blinded.
  Arms: Cohort 10^9
Biological: Placebo (for Cohort 10^8) — Gauze pads will be saturated with Placebo and then applied to each subject's volar forearm and covered with occlusive dressing once daily for 3 consecutive days. Placement of the gauze to each subject's right or left volar forearm will be randomized and double-blinded.
  Arms: Cohort 10^8
Biological: Placebo (for Cohort 10^9) — Gauze pads will be saturated with Placebo and then applied to each subject's volar forearm and covered with occlusive dressing once daily for 3 consecutive days. Placement of the gauze to each subject's right or left volar forearm will be randomized and double-blinded.
  Arms: Cohort 10^9

SUMMARY:
This study will examine the safety of ascending doses of AB-SA01 when topically applied to intact skin of healthy adults.

DETAILED DESCRIPTION:
AB-SA01 consists of three bacteriophages (viruses) that target Staphylococcus aureus bacteria.

The safety of AB-SA01 will be assessed when topically administered once daily to the volar aspect of the forearm at a dose of 10^8 plaque forming units (PFU) per phage for 3 consecutive days, and then at a dose of 10^9 plaque forming units (PFU) per phage for 3 consecutive days. Both AB-SA01 and placebo will be administered to each subject to provide his/her own control for evaluation of skin reactions. The right or left placement of the placebo will be randomized and double-blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 60 years of age, inclusive, at the time of the first treatment
2. Willing and able to sign the informed consent and adhere to the study schedule
3. Healthy subject as determined by the principal investigator or designee via medical history and clinical examination before enrollment in the study
4. Normal skin of the volar aspect of the forearms, as determined by the principal investigator or designee via examination
5. If female, the subject is not pregnant or breastfeeding and has a negative urine pregnancy test at screening, and prior to receiving the first study treatment
6. If female of childbearing potential, the subject agrees to use adequate contraception from screening, throughout the study period, and for 30 days after completion of treatment.
7. If male, subjects with female partners of childbearing potential must agree to use adequate contraception from screening, throughout the study period, and for 30 days after completion of treatment

Exclusion Criteria:

1. Any past use of a bacteriophage product, or planned use from the time of screening and during the entire study period
2. Planned participation in another clinical trial and/or use of any product that is investigational, drug, biologic or device, within 30 days preceding screening and during the entire study period
3. Skin lesions, chronic skin conditions, scars or tattoo placement, as established by skin examination before enrollment in the study that would interfere with study treatment.
4. Chronic administration (defined as more than 14 days total in the past 6 months) of immunosuppressant or other immune-modifying drugs within 6 months prior to the first study treatment
5. Chronic administration of topical steroids to the volar aspect of the forearms (defined as more than 14 days total in the 6 months prior to the first study treatment)
6. Any other prohibited medication or treatment
7. Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history, physical examination, and screening serology (HIV, HbsAg, and anti-HCV)
8. History of congenital or hereditary immunodeficiency
9. History of any severe allergic reaction or hypersensitivity (anaphylaxis)
10. History of allergic reaction or irritant contact dermatitis due to wound dressings (eg, adhesive tapes, bandages, gauze)
11. History of allergic reaction to castor oil
12. Acute disease and/or fever at the time of study treatment
13. Acute or chronic, clinically significant pulmonary, cardiovascular, neurologic, hepatic, or renal functional abnormality as determined by medical history, physical examination, or laboratory screening tests
14. Screening lab results with any Grade 2 or higher abnormality or clinically significant Grade 1 abnormality, as determined by the Common Terminology Criteria for Adverse Events (CTCAE).
15. Administration of immunoglobulins and/or any blood products within the 3 months preceding the first study treatment or planned administration during the study period
16. Recent (within 12 months prior to screening) history of chronic alcohol abuse, defined as a history of ethanol consumption on average > 40 g/day for women and 60 g/day for men for at least 12 months prior to Baseline.
17. Recent (within 12 months prior to screening) history of illicit drug abuse
18. Inability to comply with study requirements and restrictions
19. Any reason, considered by the principal investigator or designee, to preclude subject involvement in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From first dose through the End of Study visit (Day 14 ± 2 days)
  Occurrence, intensity, and relationship of adverse events (AEs) from first dose through the End of Study visit
Change from Baseline in Clinical Laboratory Tests | Day 0 (pre-dose), Day 3, and Day 14 ± 2 days
  Clinical laboratory tests (hematology, chemistry, and urinalysis)
Skin Reaction Change from Baseline | Days 0, 1, and 2 (pre- and post-dose), and on Day 3, Day 7 ± 1 day, and Day 14 ± 2 days
  skin reaction assessments

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Livezey, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Clinical Trials Center, WRAIR, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided